CLINICAL TRIAL: NCT01551095
Title: Self-Propelled Percutaneous Endoscopic GastroJejunostomy (PEG-J): A Pilot Study
Brief Title: Self-Propelled Percutaneous Endoscopic GastroJejunostomy (PEG-J)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Proof of principle was achieved after inclusion of 7 patients
Sponsor: Johns Hopkins University (Other)
Collaborators: GI Supply (Other)
Responsible Party: Principal Investigator, Mouen Khashab, Assistant Professor of Medicine; Director of Therapeutic Endoscopy, Johns Hopkins University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NA_00048369
Record Dates: First submitted 2012-02-29; First posted 2012-03-12 (Estimated); Results first posted 2016-10-12 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: GERD
Keywords: PEGJ; PEG-J; percutaneous endoscopic gastrostomy; feeding tube; gastroparesis; acute pancreatitis; stroke; respiratory failure; GERD; balloon; self-propelled
MeSH Terms: conditions — Gastroesophageal Reflux; Gastroparesis; Pancreatitis; Stroke; Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PEGJ (Experimental): Patients in this arm will receive self-propelled balloon PEGJ tube.
  Interventions: Device: PEGJ tube

INTERVENTIONS:
Device: PEGJ tube — The self-propelled PEGJ feeding tube

SUMMARY:
This research is being done to study the safety of an investigational percutaneous endoscopic gastrojejunostomy (PEGJ) tube and whether the addition of a balloon on the end of the J tube prevents it from slipping back into the stomach.

DETAILED DESCRIPTION:
The word "investigational" means the PEGJ feeding tube used in this study is not approved by the U. S. Food and Drug Administration (FDA) and is still being tested in research studies. Currently commercially available PEGJ tubes are long tubes which are placed into the part of the small intestine that connects to the stomach (duodenum) under endoscopic guidance. The tip of these PEGJ tubes usually have some built-in extra weight (several grams), which theoretically should prevent slippage of the tube back into the stomach. However, these tubes usually cannot be placed very far into the duodenum and the build-in weight is usually not sufficient to keep the tube in place.

The tip of the currently commercially available PEGJ tubes often (usually within 1-2 weeks) migrates back into the stomach and at that point the tube needs to be replaced. The investigational PEGJ feeding tube used in this study is self-propelled and has a balloon on its tip. The tip of this tube is directed endoscopically through the part of the stomach that connects to the duodenum (pylorus), then the balloon is filled with 5 cc of water and the endoscope is removed. The water filled balloon then is carried by the movement of the intestinal muscles through the duodenum into the middle section of the small intestine (jejunum). It is hoped that such a deep position of the tip of the self-propelled PEGJ tube and presence of the water-filled balloon on its tip will prevent migration of the tube back into the stomach and therefore eliminates the need for tube replacement.

The only difference between the currently approved PEGJ feeding tube and the investigational one being used in this study is the addition of the balloon to the tip of the J port. People who come to Johns Hopkins Hospital for PEGJ placement as part of standard clinical care and who are not pregnant may join the study.

ELIGIBILITY:
Inclusion Criteria:

* age 18-90 years
* need for post-pyloric feeding (patients unable to eat due to stroke, intubated patients with respiratory failure, patients with acute pancreatitis, etc)
* ability to give informed consent for the study

Exclusion Criteria:

* patients with uncorrectable bleeding disorders (INR more than 1.5, platelet count less than 50,000)
* inability to get informed consent for the study from patients or their families
* pregnancy (all women of child-bearing age will undergo urine pregnancy testing)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mouen Khashab, MD, Principal Investigator — Johns Hopkins Hospital Department of Gastroenterology
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Kim KJ, Victor D, Stein E, Valeshabad AK, Saxena P, Singh VK, Lennon AM, Clarke JO, Khashab MA. A novel ballooned-tip percutaneous endoscopic gastrojejunostomy tube: a pilot study. Gastrointest Endosc. 2013 Jul;78(1):154-7. doi: 10.1016/j.gie.2013.03.005. Epub 2013 Apr 24. PMID 23622977

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between January 2012 and May 2012 in a tertiary academic center
Period: Overall Study
Arm/Group | PEGJ
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PEGJ
Number analyzed (Participants) | 7
Age, Customized [Mean (Full Range); unit: years] | 38.3 [24 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety: Number of Participants With Adverse Events
Description: One week after the procedure patients were called by one of the study investigators and were asked whether or not they had Abdominal pain, Nausea or Vomiting after the procedure.
Time Frame: From date of PEGJ placement up to 3 weeks
Measure: Number; unit: participants
Arm/Group | PEGJ
Number analyzed (Participants) | 7
participants
  Nausea | 0
  Vomiting | 0
  Abdominal Pain | 1

2. Secondary Outcome: Number of Participants With Retrograde Migration of PEGJ Feeding Tube Within 3 Weeks of Placement
Description: An Abdominal X-ray was obtained 3 weeks after the procedure to check whether or not there was any PEGJ feeding tube migration.
Time Frame: From date of PEGJ placement up to 3 weeks
Measure: Number; unit: participants
Arm/Group | PEGJ
Number analyzed (Participants) | 7
participants | 0

ADVERSE EVENTS:
Arm/Group | PEGJ
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEGJ (N=7)
Abdominal pain (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Small number of patients and short follow-up

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No